CLINICAL TRIAL: NCT04456920
Title: Pain Monitoring After Breast Biopsy: Benefit of E-health
Acronym: BIO-PSY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PROICM 2020-06 BIO
Record Dates: First submitted 2020-06-23; First posted 2020-07-07 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Biopsy Wound
MeSH Terms: conditions — Breast Neoplasms | interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (Experimental): PRO (Patient Reported Outcomes) gathered via a phone consultation
  Interventions: Other: phone consultation; Other: visit
- Experimental group 2 (Experimental): e-PRO self-completed via connected objects (tablet/phone)
  Interventions: Other: e-PRO self-completed via connected objects (tablet/phone); Other: phone consultation; Other: visit
- Control group (No Intervention): group without e-PROs (standard care)

INTERVENTIONS:
Other: phone consultation — At D1, D2 and D3, patients in the experimental group 1 will receive a call from a neuro-psychologist during which pain, anxiety and esthetical biopsy impact will be assessed using numeric or visual analog scales during a semi-direct interview. During this call, any adverse events related to the breast biopsy will also be noted, as well as the amount, nature and dose of analgesics, anxiolytics, anti-depressants, anti-inflammatory and hypnotics taken linked to the biopsy. If detected, pain or significative distress would be specifically managed.
  Arms: Experimental group 1
Other: e-PRO self-completed via connected objects (tablet/phone) — Patients in the experimental group 2 will be asked by SMS or notification to connect to the application in order to complete online the numeric and visual anog scales of pain, anxiety and esthetical impact. Any adverse events related to the breast biopsy will also be noted online, as well as the amount, nature and dose of analgesics, anxiolytics, anti-depressants, anti-inflammatory and hypnotics taken for the biopsy. If detected, pain or significative distress would be specifically managed
  Arms: Experimental group 2
Other: phone consultation — At D4 post biopsy, all patients (of the 3 groups) will receive a phone call from a neuro-psychologist to assess pain, anxiety and esthetical impact, using numeric scales, and to collect adverse events. If detected, pain or significative distress would be specifically managed.
  Arms: Experimental group 1; Experimental group 2
Other: visit — And at D10 (+/- 2 days), all patients will physically come to the Cancer center in the consultation of biopsy results announcement. At the beginning of this consultation, pain, anxiety and esthetical impact will be assessed using numeric scales. . The adverse events related to the breast biopsy will be collected as well as the amount, nature and dose of analgesics, anxiolytics, anti-depressants, anti-inflammatory and hypnotics taken for the biopsy and its findings. Insomnia will be evaluated by the Insomnia Severity Index. If detected, pain or significative distress would be managed as usually in the center.
  Arms: Experimental group 1; Experimental group 2

SUMMARY:
Each year, approximately 1500 breast biopsies (1000 microbiopsies and 500 macrobiopsies) are performed in the radiologic department of the Montpellier Cancer Institute (ICM). This exam, which is relatively easy for the radiologist, can however lead to major anxiety for patients. Indeed, previous studies show that about 50% of women undergoing a breast biopsy have significant anxiety affects.

Anxiety associated with the risks of biopsy, potential breast cancer diagnosis and/or lack of routine sedation procedures increase patient concerns. Distress prior to biopsy is associated with greater pain and discomfort during the procedure. The psychological distress that persists after the biopsy is related to a worse psychological management of side effects of the biopsy breast (e.g., sensitivity, skin irritation).

Limiting apprehension, worry and anxiety induced by the uncertainty linked to the biopsy results and the biopsy-related pain should be an integral part of the medical care through the patient follow-up during, after and until the diagnosis is announced. In light of these challenges, new alternative methods are emerging to enhance patient knowledge, develop procedural skills, improve confidence and mitigate procedural anxiety. However, to our knowledge, few methods have been developed during this period of 'waiting-time'. Currently, only care instructions and a consultation to announce the results (about 10 days after the procedure) are proposed to patients at the end of biopsy. Patients are also encouraged to call if they suspect complications such as infection or bleeding.

In this context, the investigators propose to integrate a pain management after biopsy via e-health system through the patient's medical care. Radiologist/patient communication could have an impact on patients' anxiety and health-related issues, given the challenging nature of discussions around need for breast biopsy and potential implications of the results. Indeed, paying attention and focusing on symptoms as patients experience them improves their empowerment and their adjustment to the disease.

Web-based systems that can provide electronic-Patient reported Outcomes (e-PRO) have been shown to prompt clinicians to intensify symptom management, to improve symptom control and to enhance patient-clinician communication patient satisfaction, as well as well-being. In addition, it is known that improved communication between patients and medical staff to less anxiety after a biopsy and that anxiety is related to pain.

Taken as a whole, these elements encourage the integration of e-health and e-PRO for the management of pain and anxiety in patients undergoing a biopsy. The benefits of e-PRO are still being discussed in terms of quality of life (Qol) and psychological distress. The investigator propose to integrate two types of e-health intervention: 1/e-PRO collected by connected objects (smartphone or tablet) as they were used in previous studies, and 2/ e-PRO collected by a phone consultation, which values human communication between the medical staff and the patient.

In case of significant pain, the collection of e-PRO by any of these e-health interventions will generate an alert and a reactive and responsive care.

In fine, the purpose of this research is to improve the medical organization and care of post-biopsy patients by proposing an innovative connected patient technology, regardless of their remoteness from the hospital.

Social inequalities will be reduced by lending a tablet to patients who do not have such a device with a 4G key.

DETAILED DESCRIPTION:
The primary objective is to compare the benefit of intervention by e-health (phone consultation with a professional or connected objects (smartphone or tablet)) with the standard follow up of the pain intensity of patients 4 days (D4) after un breast biopsy.

This study is a Monocentric, prospective, open-labeled, randomized controlled trial. A total of 192 patients (64 patients in group control vs 64 patients in experimental group 1 (PRO gathered via a phone consultation) and 64 patients in experimental group 2 (e-PRO self-completed via connected objects (tablet/phone) will be required including 10% of lost-to-follow-up patients.

The inclusion period would be 8 months

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnostic breast biopsy at ICM
* Age > 18 years
* Informed patient and signed informed consent received
* Affiliation to a social security system

Exclusion Criteria:

* Patient without phone number
* Patient with previous biopsy in 6 months prior to study
* Pregnant and breastfeeding woman
* Patient whose regular follow-up is initially impossible for psychological, family, social or geographical reasons
* Patient under legal protection (guardianship, curatorship or safeguarding of justice)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nougaret Stéphanie, MD, Study Chair — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (1):
- Icm Val D'Aurelle, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients All participant data collected during the trial, after encoding with an inclusion number, 1st letter of the name and surname may be shared.
  The data of the participants will be available upon request and with the completion of a contract between the promoter and the applicant.
  The study protocol, the statistical analysis plan (PAS) and the analytical code may also be subject to data sharing as part of a transfer contract (RGPD)

REFERENCES:
- [Background] Pineault P. Breast Cancer Screening: Women's Experiences of Waiting for Further Testing. Oncol Nurs Forum. 2007 Jul;34(4):847-53. doi: 10.1188/07.ONF.847-853. PMID 17723985
- [Background] Lampic C, Thurfjell E, Bergh J, Sjoden PO. Short- and long-term anxiety and depression in women recalled after breast cancer screening. Eur J Cancer. 2001 Mar;37(4):463-9. doi: 10.1016/s0959-8049(00)00426-3. PMID 11267855
- [Background] Iwamitsu Y, Shimoda K, Abe H, Tani T, Okawa M, Buck R. Anxiety, emotional suppression, and psychological distress before and after breast cancer diagnosis. Psychosomatics. 2005 Jan-Feb;46(1):19-24. doi: 10.1176/appi.psy.46.1.19. PMID 15765817
- [Background] Grimm LJ, Shelby RA, Knippa EE, Langman EL, Miller LS, Whiteside BE, Soo MSC. Patient Perceptions of Breast Cancer Risk in Imaging-Detected Low-Risk Scenarios and Thresholds for Desired Intervention: A Multi-Institution Survey. J Am Coll Radiol. 2018 Jun;15(6):911-919. doi: 10.1016/j.jacr.2018.02.010. Epub 2018 Mar 30. PMID 29606632
- [Background] Dorfman CS, Lamb E, Van Denburg A, Wren AA, Soo MS, Faircloth K, Gandhi V, Shelby RA. The relationship between holding back from communicating about breast concerns and anxiety in the year following breast biopsy. J Psychosoc Oncol. 2018 Mar-Apr;36(2):222-237. doi: 10.1080/07347332.2017.1395939. Epub 2018 Jan 11. PMID 29064780
- [Background] Andrykowski MA, Carpenter JS, Studts JL, Cordova MJ, Cunningham LL, Beacham A, Sloan D, Kenady D, McGrath P. Psychological impact of benign breast biopsy: a longitudinal, comparative study. Health Psychol. 2002 Sep;21(5):485-94. PMID 12211516
- [Background] Mema E, Cho E, Ryu YK, Jadeja P, Wynn R, Taback B, Ha R. In the Setting of Negative Mammogram, Is Additional Breast Ultrasound Necessary for Evaluation of Breast Pain? Curr Probl Diagn Radiol. 2019 Mar-Apr;48(2):117-120. doi: 10.1067/j.cpradiol.2017.12.007. Epub 2018 Jan 9. PMID 29402490
- [Background] Roark AA, Ebuoma LO, Ortiz-Perez T, Sepulveda KA, Severs FJ, Wang T, Benveniste AP, Sedgwick EL. Impact of Simulation-Based Training on Radiology Trainee Education in Ultrasound-Guided Breast Biopsies. J Am Coll Radiol. 2018 Oct;15(10):1458-1463. doi: 10.1016/j.jacr.2017.09.016. Epub 2017 Dec 6. PMID 29222002
- [Background] Denis F, Lethrosne C, Pourel N, Molinier O, Pointreau Y, Domont J, Bourgeois H, Senellart H, Tremolieres P, Lizee T, Bennouna J, Urban T, El Khouri C, Charron A, Septans AL, Balavoine M, Landry S, Solal-Celigny P, Letellier C. Randomized Trial Comparing a Web-Mediated Follow-up With Routine Surveillance in Lung Cancer Patients. J Natl Cancer Inst. 2017 Sep 1;109(9). doi: 10.1093/jnci/djx029. PMID 28423407
- [Background] Basch E, Artz D, Dulko D, Scher K, Sabbatini P, Hensley M, Mitra N, Speakman J, McCabe M, Schrag D. Patient online self-reporting of toxicity symptoms during chemotherapy. J Clin Oncol. 2005 May 20;23(15):3552-61. doi: 10.1200/JCO.2005.04.275. PMID 15908666
- [Background] Berry DL, Blumenstein BA, Halpenny B, Wolpin S, Fann JR, Austin-Seymour M, Bush N, Karras BT, Lober WB, McCorkle R. Enhancing patient-provider communication with the electronic self-report assessment for cancer: a randomized trial. J Clin Oncol. 2011 Mar 10;29(8):1029-35. doi: 10.1200/JCO.2010.30.3909. Epub 2011 Jan 31. PMID 21282548
- [Background] Chen J, Ou L, Hollis SJ. A systematic review of the impact of routine collection of patient reported outcome measures on patients, providers and health organisations in an oncologic setting. BMC Health Serv Res. 2013 Jun 11;13:211. doi: 10.1186/1472-6963-13-211. PMID 23758898
- [Background] Detmar SB, Muller MJ, Schornagel JH, Wever LD, Aaronson NK. Health-related quality-of-life assessments and patient-physician communication: a randomized controlled trial. JAMA. 2002 Dec 18;288(23):3027-34. doi: 10.1001/jama.288.23.3027. PMID 12479768
- [Background] Kotronoulas G, Kearney N, Maguire R, Harrow A, Di Domenico D, Croy S, MacGillivray S. What is the value of the routine use of patient-reported outcome measures toward improvement of patient outcomes, processes of care, and health service outcomes in cancer care? A systematic review of controlled trials. J Clin Oncol. 2014 May 10;32(14):1480-501. doi: 10.1200/JCO.2013.53.5948. Epub 2014 Apr 7. PMID 24711559
- [Background] Valderas JM, Kotzeva A, Espallargues M, Guyatt G, Ferrans CE, Halyard MY, Revicki DA, Symonds T, Parada A, Alonso J. The impact of measuring patient-reported outcomes in clinical practice: a systematic review of the literature. Qual Life Res. 2008 Mar;17(2):179-93. doi: 10.1007/s11136-007-9295-0. Epub 2008 Jan 4. PMID 18175207
- [Background] Velikova G, Booth L, Smith AB, Brown PM, Lynch P, Brown JM, Selby PJ. Measuring quality of life in routine oncology practice improves communication and patient well-being: a randomized controlled trial. J Clin Oncol. 2004 Feb 15;22(4):714-24. doi: 10.1200/JCO.2004.06.078. PMID 14966096
- [Background] Kroenke K, Krebs EE, Wu J, Yu Z, Chumbler NR, Bair MJ. Telecare collaborative management of chronic pain in primary care: a randomized clinical trial. JAMA. 2014 Jul 16;312(3):240-8. doi: 10.1001/jama.2014.7689. PMID 25027139
- [Background] Santana MJ, Feeny D, Johnson JA, McAlister FA, Kim D, Weinkauf J, Lien DC. Assessing the use of health-related quality of life measures in the routine clinical care of lung-transplant patients. Qual Life Res. 2010 Apr;19(3):371-9. doi: 10.1007/s11136-010-9599-3. Epub 2010 Feb 10. PMID 20146009
- [Background] Seow H, Sussman J, Martelli-Reid L, Pond G, Bainbridge D. Do high symptom scores trigger clinical actions? An audit after implementing electronic symptom screening. J Oncol Pract. 2012 Nov;8(6):e142-8. doi: 10.1200/JOP.2011.000525. Epub 2012 Aug 21. PMID 23598849
- [Background] Atkinson TM, Ryan SJ, Bennett AV, Stover AM, Saracino RM, Rogak LJ, Jewell ST, Matsoukas K, Li Y, Basch E. The association between clinician-based common terminology criteria for adverse events (CTCAE) and patient-reported outcomes (PRO): a systematic review. Support Care Cancer. 2016 Aug;24(8):3669-76. doi: 10.1007/s00520-016-3297-9. Epub 2016 Jun 3. PMID 27260018
- [Background] Miller LS, Shelby RA, Balmadrid MH, Yoon S, Baker JA, Wildermann L, Soo MS. Patient anxiety before and immediately after imaging-guided breast biopsy procedures: impact of radiologist-patient communication. J Am Coll Radiol. 2013 Jun;10(6):423-31. doi: 10.1016/j.jacr.2012.11.005. Epub 2013 Mar 15. PMID 23499400
- [Background] Aitken RC. Measurement of feelings using visual analogue scales. Proc R Soc Med. 1969 Oct;62(10):989-93. doi: 10.1177/003591576906201005. No abstract available. PMID 4899510
- [Background] Hjermstad MJ, Fayers PM, Haugen DF, Caraceni A, Hanks GW, Loge JH, Fainsinger R, Aass N, Kaasa S; European Palliative Care Research Collaborative (EPCRC). Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage. 2011 Jun;41(6):1073-93. doi: 10.1016/j.jpainsymman.2010.08.016. PMID 21621130
- [Background] Wilkie D, Lovejoy N, Dodd M, Tesler M. Cancer pain intensity measurement: concurrent validity of three tools--finger dynamometer, pain intensity number scale, visual analogue scale. Hosp J. 1990;6(1):1-13. doi: 10.1080/0742-969x.1990.11882662. PMID 2379920
- [Background] Chen PY, Yang CM, Morin CM. Validating the cross-cultural factor structure and invariance property of the Insomnia Severity Index: evidence based on ordinal EFA and CFA. Sleep Med. 2015 May;16(5):598-603. doi: 10.1016/j.sleep.2014.11.016. Epub 2015 Feb 12. PMID 25863811
- [Background] Elkins G, Staniunas R, Rajab MH, Marcus J, Snyder T. Use of a numeric visual analog anxiety scale among patients undergoing colorectal surgery. Clin Nurs Res. 2004 Aug;13(3):237-44. doi: 10.1177/1054773803262222. PMID 15245638
- [Background] Hodkinson B, Maheu E, Michon M, Carrat F, Berenbaum F. Assessment and determinants of aesthetic discomfort in hand osteoarthritis. Ann Rheum Dis. 2012 Jan;71(1):45-9. doi: 10.1136/ard.2011.153965. Epub 2011 Sep 6. PMID 21900283
- [Background] Yennurajalingam S, Kang JH, Hui D, Kang DH, Kim SH, Bruera E. Clinical response to an outpatient palliative care consultation in patients with advanced cancer and cancer pain. J Pain Symptom Manage. 2012 Sep;44(3):340-50. doi: 10.1016/j.jpainsymman.2011.09.014. Epub 2012 Jun 13. PMID 22699092
- [Background] den Heijer M, Seynaeve C, Vanheusden K, Duivenvoorden HJ, Bartels CC, Menke-Pluymers MB, Tibben A. Psychological distress in women at risk for hereditary breast cancer: the role of family communication and perceived social support. Psychooncology. 2011 Dec;20(12):1317-23. doi: 10.1002/pon.1850. Epub 2010 Oct 5. PMID 20925135
- [Background] Manne S, Myers S, Ozga M, Kissane D, Kashy D, Rubin S, Heckman C, Rosenblum N. Holding back sharing concerns, dispositional emotional expressivity, perceived unsupportive responses and distress among women newly diagnosed with gynecological cancers. Gen Hosp Psychiatry. 2014 Jan-Feb;36(1):81-7. doi: 10.1016/j.genhosppsych.2013.10.001. Epub 2013 Oct 9. PMID 24211156
- [Background] Cordova MJ, Cunningham LL, Carlson CR, Andrykowski MA. Social constraints, cognitive processing, and adjustment to breast cancer. J Consult Clin Psychol. 2001 Aug;69(4):706-11. PMID 11550737

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Group 1: PRO (Patient Reported Outcomes) gathered via a phone consultation
  phone consultation: At D1, D2 and D3, patients in the experimental group 1 will receive a call from a neuro-psychologist during which pain, anxiety and esthetical biopsy impact will be assessed using numeric or visual analog scales during a semi-direct interview. During this call, any adverse events related to the breast biopsy and concomitant treatment taken will be collected. If detected, pain or significative distress would be specifically managed.
  phone consultation: At D4 post biopsy, patients will receive a phone call from a neuro-psychologist to assess pain, anxiety and esthetical impact, using numeric scales, and to collect adverse events. If detected, pain or significative distress would be specifically managed.
  visit: And at D10 (+/- 2 days), all patients will physically come to the Cancer center in the consultation of biopsy results announcement. At the beginning of this consultation, pain, anxiety and esthetical impact will be assessed using numeric scales. . The adverse events related to the breast biopsy and concomitant treatment taken will be collected. Insomnia will be evaluated by the Insomnia Severity Index. If detected, pain or significative distress would be managed as usually in the center.
- Experimental Group 2: e-PRO self-completed via connected objects (tablet/phone)
  e-PRO self-completed via connected objects (tablet/phone): Patients in the experimental group 2 will be asked by SMS or notification to connect to the application in order to complete online the numeric and visual anog scales of pain, anxiety and esthetical impact. Any adverse events related to the breast biopsy will also be noted online, as well as concomitant treatment taken. If detected, pain or significative distress would be specifically managed
  phone consultation: At D4 post biopsy, all patients (of the 3 groups) will receive a phone call from a neuro-psychologist to assess pain, anxiety and esthetical impact, using numeric scales, and to collect adverse events. If detected, pain or significative distress would be specifically managed.
  And at D10 (+/- 2 days), all patients will physically come to the Cancer center in the consultation of biopsy results announcement. At the beginning of this consultation, pain, anxiety and esthetical impact will be assessed using numeric scales. . The adverse events related to the breast biopsy and concomitant treatment taken will be collected. Insomnia will be evaluated by the Insomnia Severity Index. If detected, pain or significative distress would be managed as usually in the center.
Period: Overall Study
Arm/Group | Experimental Group 1 | Experimental Group 2 | Control Group
Started | 63 | 65 | 65
Completed | 63 | 65 | 65
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: patients were randomized to the following stratification factors:
  * Ultrasound-guided biopsy (Microbiopsies) versus stereotactic biopsy/MRI (macrobiopsies)
  * ACR3 vs. ACR 4-5
  * Pain < 4 versus 4 at inclusion
Groups:
- Experimental Group 1: PRO (Patient Reported Outcomes) gathered via a phone consultation
  phone consultation: At D1, D2 and D3, patients in the experimental group 1 will receive a call from a neuro-psychologist during which pain, anxiety and esthetical biopsy impact will be assessed using numeric or visual analog scales during a semi-direct interview. During this call, any adverse events related to the breast biopsy and concomitant treatment taken will be collected. If detected, pain or significative distress would be specifically managed.
  phone consultation: At D4 post biopsy, patients will receive a phone call from a neuro-psychologist to assess pain, anxiety and esthetical impact, using numeric scales, and to collect adverse events. If detected, pain or significative distress would be specifically managed.
  And at D10 (+/- 2 days), all patients will physically come to the Cancer center in the consultation of biopsy results announcement. At the beginning of this consultation, pain, anxiety and esthetical impact will be assessed using numeric scales. . The adverse events related to the breast biopsy and concomitant treatment taken will be collected. Insomnia will be evaluated by the Insomnia Severity Index. If detected, pain or significative distress would be managed as usually in the center.
- Total: Total of all reporting groups
Arm/Group | Experimental Group 1 | Experimental Group 2 | Control Group | Total
Number analyzed (Participants) | 63 | 65 | 65 | 193
Age, Continuous [Median (Full Range); unit: years] | 52 [22 to 85] | 55 [22 to 82] | 56 [41 to 81] | 54 [22 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 65 | 65 | 193
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Type of biopsy [Count of Participants; unit: Participants]
  Macrobiopsy | 42 | 43 | 42 | 127
  Microbiopsy | 21 | 22 | 23 | 66
ACR [Number; unit: participants]
  Grade 3 of ACR (American College of Radiology) better outcome | 0 | 3 | 2 | 5
  Grade 4-5 of ACR (American College of Radiology worse outcomes | 63 | 62 | 63 | 188
Pain at the baseline [Number; unit: participants]
  Pain Score < 4 on a numeric pain scale (from 0 to 10) | 50 | 51 | 51 | 152
  Pain Score >= 4 on a numeric pain scale (from 0 to 10) | 13 | 14 | 14 | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants by Pain Intensity at Day 4 Post Breast Biopsy With a Benefit of Intervention by E-health (Phone Consultation With a Professional or Connected Objects (Smartphone or Tablet)) Compared of the Standard Follow up
Description: Pain score assessed (by phone) via a numeric pain scale (from 0 "no pain" to 10 "maximal pain")completed 4 days after biopsy (Day 4).
Time Frame: From date of randomization until the Day 4 post biopsy
Measure: Number; unit: participants
Arm/Group | Experimental Group 1 | Experimental Group 2 | Control Group
Number analyzed (Participants) | 58 | 61 | 60
participants
  No pain (0) on a a numeric pain scale | 39 | 43 | 36
  Low pain score (1 to 3) on a a numeric pain scale | 19 | 17 | 22
  Moderate pain Score (4 to 5) on a a numeric pain scale | 0 | 1 | 1
  Intense pain Score (6 to 7) on a a numeric pain scale | 0 | 0 | 1

2. Secondary Outcome: Pain Intensity During the Consultation of Results Announcement After a Breast Biopsy Between the Benefit of Intervention by E-health (Phone Consultation With a Professional or Connected Objects) Compared to the Standard Follow up
Description: Pain score assessed using a numeric pain scale (from 0 "no pain" to 10 "maximal pain") administered after to biopsy and during the consultation of results announcement (approximately Day 10).
Time Frame: From date of randomization until the Day 10 post biopsy
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Experimental Group 1 | Experimental Group 2 | Control Group
Number analyzed (Participants) | 63 | 65 | 65
score on a scale
  Pain score (0,10) at J0 on a numeric pain scale | 1 [0 to 8] | 1 [0 to 9] | 1 [0 to 9]
  Pain score (0,10) at J10 on a numeric pain scale | 0 [0 to 5] | 0 [0 to 4] | 0 [0 to 5]

3. Secondary Outcome: the Benefit According to the Type of Intervention by E-health (Phone Consultation With a Professional or Connected Objects) on the Pain Intensity of Patients at 4 Days (D4) and During the Consultation of Results Announcement After a Breast Biopsy.
Description: Pain score assessed using a numeric pain scale (from 0 "no pain" to 10 "maximal pain") administered after to biopsy, at 4 days and 10 days post biopsy
Time Frame: From date of randomization until the Day 4 / Day 10 post biopsy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group 1 | Experimental Group 2 | Control Group
Number analyzed (Participants) | 63 | 65 | 65
score on a scale
  Pain score (from 0 to10) at biopsy day on a numeric pain scale | 2.08 (2.50) | 1.98 (2.21) | 1.86 (1.78)
  Pain score (from 0 to 10) Day 4 post biopsy on a numeric pain scale | 0.47 (0.78) | 0.54 (1.03) | 0.65 (1.12)
  Pain score (from 0 to 10) Day 10 post biopsy on a numeric pain scale | 0.75 (1.35) | 0.54 (1.10) | 0.54 (0.99)

4. Secondary Outcome: the Benefit of Intervention by E-health (Phone Consultation With a Professional or Connected Objects) With the Standard Follow up of the Anxiety Intensity of Patients at 4 Days and During the Consultation of Results Announcement, After a Breast Biopsy.
Description: Anxiety score assessed using a numeric anxiety scale (from 0 "no anxiety" to 10 "maximal anxiety") administered after to biopsy, at 4 days (Day 4) and 10 days (Day 10)
Time Frame: From date of randomization until the Day 4 and Day 10 post biopsy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group 1 | Experimental Group 2 | Control Group
Number analyzed (Participants) | 63 | 65 | 65
score on a scale
  Anxiety score (0,10) at J0 on a numeric anxiety scale | 4.52 (3.02) | 4.12 (3.31) | 4.57 (3.27)
  Anxiety score (0,10) at J4 a numeric anxiety scale | 1.88 (1.63) | 2.51 (2.75) | 3.80 (2.50)
  Anxiety score (0,10) at J10 a numeric anxiety scale | 3.43 (3.02) | 3.83 (3.00) | 4.65 (3.19)

5. Secondary Outcome: the Benefit of Intervention by E-health (Phone Consultation With a Professional or Connected Objects) With the Standard Follow up of the Esthetic Impact of Patients at 4 and 10 Days (D4, D10) After a Breast Biopsy.
Description: Esthetic impact score assessed using a numeric esthetic scale (from 0 "no impact" to 100 "maximal impact") administered after to biopsy, at 4 days and 10 days post biopsy
Time Frame: From date of randomization until the Day 4 and Day 10 post biopsy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group 1 | Experimental Group 2 | Control Group
Number analyzed (Participants) | 63 | 65 | 65
score on a scale
  Esthetic Impact (0-100) at J0 on a numeric scale | 4.29 (10.88) | 4.06 (8.49) | 6.41 (12.77)
  Esthetic Impact (0-100) at J4 on a numeric scale | 7.69 (19.00) | 10.05 (21.77) | 4.18 (8.43)
  Esthetic Impact (0-100) at J10 on a numeric scale | 8.69 (17.08) | 8.54 (15.91) | 3.08 (5.84)

6. Secondary Outcome: the Benefit According to the Type of Intervention by E-health (Phone Consultation With a Professional or Connected Objects) on the Insomnia of Patients at 10 Days (About Day 10), After a Breast Biopsy.
Description: Insomnia score assessed using the Index of Severity of Insomnia (from 0 "no insomnia" to 28 "maximal insomnia") administered at 10 days post biopsy
Time Frame: From date of randomization until the Day 10 post biopsy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group 1 | Experimental Group 2 | Control Group
Number analyzed (Participants) | 63 | 65 | 65
score on a scale
  Insomnia score (0 to 28) at J0 | 7.88 (5.90) | 7.42 (5.97) | 7.22 (5.57)
  Insomnia score (0 to 28) at J10 | 7.43 (6.43) | 6.65 (5.95) | 7.34 (5.91)

7. Secondary Outcome: the Benefit of Intervention by E-health (Phone Consultation With a Professional or Connected Objects) With the Standard Follow up of Patient's Management
Description: Number of alerts that generated a phone call or number of phone calls generated directly by the patient and patient care accordingly.
Time Frame: From date of randomization until the Day 4 and the Day 10 post biopsy
Measure: Number; unit: participants
Arm/Group | Experimental Group 1 | Experimental Group 2 | Control Group
Number analyzed (Participants) | 63 | 65 | 65
participants
  Phone call | 60 | 62 | 62
  No phone call | 0 | 1 | 0
  No data | 3 | 2 | 3

8. Secondary Outcome: the Use of a Biopsy-related Drug Intervention in Patients With E-health Interventions (Phone Consultation or Smartphone), With the Standard Follow-up, at 10 Days After a Breast Biopsy.
Description: Quantity, nature and dose of treatments used for the biopsy and its aftermath.
Time Frame: From date of randomization until the Day 4 and Day 10 post biopsy
Measure: Number; unit: participants
Arm/Group | Experimental Group 1 | Experimental Group 2 | Control Group
Number analyzed (Participants) | 63 | 65 | 65
participants
  concomitant treatment | 23 | 28 | 27
  No concomitant treatment | 40 | 36 | 38
  No data | 0 | 1 | 0

9. Secondary Outcome: Adverse Events in Patients With E-health Interventions (Phone Consultation With a Professional or Connected Objects), With the Standard Follow-up, During the Consultation of Results Announcement (About D10) After a Breast Biopsy.
Description: Adverse event in particular bleeding and infection due to biopsy recorded at 4 days (Day 4) and during the consultation of results announcement (about Day 10) by NCI-CTCAE 5.0
Time Frame: From date of randomization until the Day 4 and the Day 10 post biopsy
Measure: Number; unit: participants
Arm/Group | Experimental Group 1 | Experimental Group 2 | Control Group
Number analyzed (Participants) | 63 | 65 | 65
participants
  Bleeding | 0 | 1 | 1
  no bleeding | 63 | 64 | 64
  Infection | 0 | 0 | 0
  no infection | 63 | 65 | 65

10. Secondary Outcome: Assess Satisfaction With Specific Study Management.
Description: Number of positive responses to satisfaction questions (from 0 (no satisfy) to 10 (veryy satisfy) related to the number of solicitations for the study and how interventions are communicated.
  No response 1, 2, 3, 4, 5, and 6 done.
Time Frame: at the Day 10 post biopsy
Measure: Number; unit: participants
Groups:
- Experimental Group 2: e-PRO (Patient Reported Outcomes) self-completed via connected objects (tablet/phone)
  e-PRO (Patient Reported Outcomes) self-completed via connected objects (tablet/phone): Patients in the experimental group 2 will be asked by SMS or notification to connect to the application in order to complete online the numeric and visual anog scales of pain, anxiety and esthetical impact. Any adverse events related to the breast biopsy will also be noted online, as well as concomitant treatment taken. If detected, pain or significative distress would be specifically managed
  phone consultation: At D4 post biopsy, all patients (of the 3 groups) will receive a phone call from a neuro-psychologist to assess pain, anxiety and esthetical impact, using numeric scales, and to collect adverse events. If detected, pain or significative distress would be specifically managed.
  And at D10 (+/- 2 days), all patients will physically come to the Cancer center in the consultation of biopsy results announcement. At the beginning of this consultation, pain, anxiety and esthetical impact will be assessed using numeric scales. . The adverse events related to the breast biopsy and concomitant treatment taken will be collected. Insomnia will be evaluated by the Insomnia Severity Index. If detected, pain or significative distress would be managed as usually in the center.
- Control Group: group without e-PROs (Patient Reported Outcomes) (standard care)
Arm/Group | Experimental Group 1 | Experimental Group 2 | Control Group
Number analyzed (Participants) | 63 | 65 | 65
participants
  7 on a numeric scale (from 0 to 10) | 2 | 1 | 1
  8 on a numeric scale (from 0 to 10) | 2 | 6 | 6
  9 on a numeric scale (from 0 to 10) | 25 | 15 | 20
  10 on a numeric scale (from 0 to 10) | 28 | 41 | 38
  no Data | 6 | 2 | 0

11. Secondary Outcome: Assess Compliance.
Description: Rate of completion questionnaire (on the application) for the patient of arm "experimental group 1" (PRO (Patient Reported Outcomes) gathered via a phone consultation). ony this arm is analysed on this secondary objective.
  indeed the objective is to evaluate compliance with an e-Health application
Time Frame: at the Day 1, 2 and 3
Population: only arm "experimental group 1" (PRO (Patient Reported Outcomes) gathered via a phone consultation) is analysed on this secondary objective other arms don't use ePRO. So this objective is only for 63 patient
Measure: Number; unit: participants
Arm/Group | Experimental Group 1
Number analyzed (Participants) | 63
participants
  completion questionnaire at Day 1 | 60
  completion questionnaire at Day 2 | 60
  completion questionnaire at DAy 3 | 59

12. Secondary Outcome: Assess Compliance.
Description: numeric scale (likert scala : (from 0 "no satisfy" to 10 "maximal satisfaction).
  no response 1, 2, 3, 4, 5 and 6
Time Frame: At the Day 3
Measure: Number; unit: participants
Arm/Group | Experimental Group 1 | Experimental Group 2 | Control Group
Number analyzed (Participants) | 63 | 65 | 65
participants
  satisfy Score 7 on a numeric scale | 2 | 1 | 1
  satisfy Score 8 on a numeric scale | 2 | 6 | 6
  satisfy Score 9 on a numeric scale | 25 | 15 | 20
  satisfy Score 10 on a numeric scale | 28 | 41 | 38
  No data | 6 | 2 | 0

ADVERSE EVENTS:
Time Frame: From randomization ti Day 10 post Biopsy
Arm/Group | Experimental Group 1 | Experimental Group 2 | Control Group
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/65 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/65 | 0/65
Other Adverse Events (participants affected / at risk) | 44/63 | 27/65 | 31/65
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group 1 (N=63) | Experimental Group 2 (N=65) | Control Group (N=65)
PAIN (General disorders) | 10 (14) | 1 (1) | 3 (4)
Anxiety (General disorders) | 23 (49) | 13 (15) | 24 (30)
Esthetic Impact (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (4) | 1 (1)
Edema (Blood and lymphatic system disorders) | 2 (3) | 2 (2) | 0 (0)
Bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Arthrophlebitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hematome (Blood and lymphatic system disorders) | 4 (12) | 6 (7) | 1 (1)
Irritation (General disorders) | 0 | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Insomnia (General disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/20/NCT04456920/Prot_SAP_000.pdf